CLINICAL TRIAL: NCT00347269
Title: Coordinated Anxiety Learning and Management (CALM): Improving Primary Care Anxiety Outcomes
Brief Title: Primary Care Intervention Strategy for Anxiety Disorders
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Peter Roy-Byrne, Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 28630; U01MH057858-05 (NIH); DSIR 83-ATAS (Other: NIMH Program Class Code)
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2017-05-19 (Actual); Last update posted 2017-05-19 (Actual); Status verified 2017-04

CONDITIONS: Post-traumatic Stress Disorder; Generalized Anxiety Disorder; Panic Disorder; Social Anxiety Disorder
Keywords: Anxiety Disorders; Post-traumatic Stress Disorder; Generalized Anxiety Disorder; Panic Disorder; Social Anxiety Disorder; Stress; Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Mental Health Disorders
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Generalized Anxiety Disorder; Panic Disorder; Phobia, Social; Anxiety Disorders; Stress Disorders, Traumatic | interventions — Cognitive Behavioral Therapy; Selective Serotonin Reuptake Inhibitors; Serotonin and Noradrenaline Reuptake Inhibitors; Benzodiazepines; Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CALM Intervention (Experimental): Participant choice of:
  Cognitive Behavioral Therapy (CBT) Psychotropic (anti-anxiety) medication optimization
  Interventions: Behavioral: Cognitive-behavioral therapy; Drug: Psychotropic medication optimization
- Treatment as Usual (TAU) (Active Comparator): Participants assigned to TAU with their primary care provider (PCP)
  Interventions: Behavioral: Treatment as Usual

INTERVENTIONS:
Behavioral: Cognitive-behavioral therapy — Participants in CALM will choose to receive CBT, medication, or both for the treatment of their anxiety. CBT includes computer-assisted CBT with an anxiety clinical specialist.
  Arms: CALM Intervention
Drug: Psychotropic medication optimization — For those participants in CALM who choose medication, the ACS will facilitate the delivery of, and adherence to, anti-anxiety medication which will be prescribed by the participants' PCP.
  Other Names: SSRI, SNRI, Benzodiazepine,
  Arms: CALM Intervention
Behavioral: Treatment as Usual — Participants in the control group will receive standard treatment from their PCP.
  Arms: Treatment as Usual (TAU)

SUMMARY:
This study will compare the effectiveness of an intervention strategy for the treatment of people with post traumatic stress disorder, generalized anxiety disorder, panic disorder, and social anxiety disorder in the primary care setting.

DETAILED DESCRIPTION:
Anxiety disorders are highly prevalent, distressing, and disabling. Most patients with anxiety disorders who do receive mental health treatment receive it in primary care settings, where the quality of care is generally insufficient. This intervention is geared towards testing the clinical effectiveness of a care-manager assisted chronic disease management program for four common anxiety disorders (post-traumatic stress disorder, generalized anxiety disorder, panic disorder, and social anxiety disorder) in the primary care setting. This approach has been shown to be effective for the treatment of depression.

Participants in this randomized, controlled trial will either be assigned to the control group: treatment-as-usual (TAU) from their primary care provider (PCP); or to the intervention group: CALM (Coordinated Anxiety Learning and Management). Intervention subjects will choose to receive CBT, medication, or both for the treatment of their anxiety. Those who choose CBT will receive it from a study-trained Anxiety Clinical Specialist (ACS) in their respective clinic. For those who choose medication, the ACS will facilitate the delivery of, and adherence to, anti-anxiety medication which will be prescribed by the participant's PCP. In this stepped-care design, subject progress will be formally re-evaluated at 8-12 week intervals. If treatment progress is not satisfactory, options include: additional or modified treatment with current modality, switching to the other treatment modality, or adding the other modality. When remission is attained, the ACS will follow-up with participants on a monthly basis to review progress and practice anxiety-reduction strategies. Treatment will continue for up to 12 months. Participants in both study arms will undergo formal baseline and outcome assessment interviews conducted at the 6, 12, and 18 month follow-up time-points.

ELIGIBILITY:
Inclusion Criteria:

* MINI diagnosed Anxiety Disorder (PTSD, GAD, SAD, PD)
* Speak English or Spanish (English only at UAMS site)

Exclusion Criteria:

* Diagnosis of Bipolar 1
* Drug and alcohol dependence; or abuse of any substance other than marijuana and alcohol
* Acute suicidality or homicidality

Eligible subjects must be current patients at one of the participating primary care clinics which include:

University of Washington:

* Harborview's Adult Medicine Clinic
* Harborview's Family Medicine Clinic
* UWMC's General Internal Medicine Clinic at Roosevelt Clinic
* PSNHC's 45th Street Clinic
* Country Doctor Community Clinic
* Carolyn Downs Family Medical Center

UCLA:

* Desert Medical Group, Palm Springs CA
* High Desert Medical Group, Lancaster, CA

UCSD:

* Kaiser Permanente, Bonita Medical Offices
* Kaiser Permanente, Otay Mesa Outpatient Medical Center
* UCSD Medical Center, Scripps Ranch Medical Office
* UCSD Medical Center, Fourth and Lewis Medical Office
* UCSD Medical Center, Perlman Ambulatory Care Center
* Sharp Rees-Stealy Medical Group, El Cajon
* Sharp Rees-Stealy Medical Group, Mira Mesa

UAMS:

* UAMS UPMG
* Little Rock Diagnostic Clinic
* St. Vincent's Family Clinic South

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1004 (Actual)
Dates: Start 2006-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter P. Roy-Byrne, MD, Principal Investigator — University of Washington; Cathy D. Sherbourne, PhD, Principal Investigator — RAND Corporation, Santa Monica, CA; Michelle G. Craske, PhD, Principal Investigator — University of California, Los Angeles; Greer Sullivan, MD, MSPH, Principal Investigator — University of Arkansas for Medical Sciences, Little Rock, AR; Murray B. Stein, MD, MPH, Principal Investigator — University of California, San Diego, San Diego, CA; Kristin Bumgardner, BS, Study Director — University of Washington
Locations (4):
- United States (4):
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - University of California, La Jolla, California
  - University of California, Los Angeles, California
  - University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Limited access datasets are available through the National Database for Clinical Trials Related to Mental Illness (NDCT), part of the NIMH Data Archive: https://data-archive.nimh.nih.gov/ndct/.

REFERENCES:
- [Background] Lang AJ, Wilkins K, Roy-Byrne PP, Golinelli D, Chavira D, Sherbourne C, Rose RD, Bystritsky A, Sullivan G, Craske MG, Stein MB. Abbreviated PTSD Checklist (PCL) as a guide to clinical response. Gen Hosp Psychiatry. 2012 Jul-Aug;34(4):332-8. doi: 10.1016/j.genhosppsych.2012.02.003. Epub 2012 Mar 27. PMID 22460001
- [Background] Craske MG, Roy-Byrne PP, Stein MB, Sullivan G, Sherbourne C, Bystritsky A. Treatment for anxiety disorders: Efficacy to effectiveness to implementation. Behav Res Ther. 2009 Nov;47(11):931-7. doi: 10.1016/j.brat.2009.07.012. Epub 2009 Jul 14. PMID 19632667
- [Background] Roy-Byrne P, Veitengruber JP, Bystritsky A, Edlund MJ, Sullivan G, Craske MG, Welch SS, Rose R, Stein MB. Brief intervention for anxiety in primary care patients. J Am Board Fam Med. 2009 Mar-Apr;22(2):175-86. doi: 10.3122/jabfm.2009.02.080078. PMID 19264941
- [Background] Campbell-Sills L, Norman SB, Craske MG, Sullivan G, Lang AJ, Chavira DA, Bystritsky A, Sherbourne C, Roy-Byrne P, Stein MB. Validation of a brief measure of anxiety-related severity and impairment: the Overall Anxiety Severity and Impairment Scale (OASIS). J Affect Disord. 2009 Jan;112(1-3):92-101. doi: 10.1016/j.jad.2008.03.014. Epub 2008 May 16. PMID 18486238
- [Background] Sullivan G, Craske MG, Sherbourne C, Edlund MJ, Rose RD, Golinelli D, Chavira DA, Bystritsky A, Stein MB, Roy-Byrne PP. Design of the Coordinated Anxiety Learning and Management (CALM) study: innovations in collaborative care for anxiety disorders. Gen Hosp Psychiatry. 2007 Sep-Oct;29(5):379-87. doi: 10.1016/j.genhosppsych.2007.04.005. PMID 17888803
- [Result] Brown LA, Krull JL, Roy-Byrne P, Sherbourne CD, Stein MB, Sullivan G, Rose RD, Bystritsky A, Craske MG. An examination of the bidirectional relationship between functioning and symptom levels in patients with anxiety disorders in the CALM study. Psychol Med. 2015 Feb;45(3):647-61. doi: 10.1017/S0033291714002062. Epub 2014 Oct 2. PMID 25272965
- [Result] Brown LA, Wiley JF, Wolitzky-Taylor K, Roy-Byrne P, Sherbourne C, Stein MB, Sullivan G, Rose RD, Bystritsky A, Craske MG. Changes in self-efficacy and outcome expectancy as predictors of anxiety outcomes from the CALM study. Depress Anxiety. 2014 Aug;31(8):678-89. doi: 10.1002/da.22256. Epub 2014 Mar 11. PMID 24619599
- [Result] Chavira DA, Golinelli D, Sherbourne C, Stein MB, Sullivan G, Bystritsky A, Rose RD, Lang AJ, Campbell-Sills L, Welch S, Bumgardner K, Glenn D, Barrios V, Roy-Byrne P, Craske M. Treatment engagement and response to CBT among Latinos with anxiety disorders in primary care. J Consult Clin Psychol. 2014 Jun;82(3):392-403. doi: 10.1037/a0036365. Epub 2014 Mar 24. PMID 24660674
- [Result] Dour HJ, Wiley JF, Roy-Byrne P, Stein MB, Sullivan G, Sherbourne CD, Bystritsky A, Rose RD, Craske MG. Perceived social support mediates anxiety and depressive symptom changes following primary care intervention. Depress Anxiety. 2014 May;31(5):436-42. doi: 10.1002/da.22216. Epub 2013 Dec 12. PMID 24338947
- [Result] Joesch JM, Golinelli D, Sherbourne CD, Sullivan G, Stein MB, Craske MG, Roy-Byrne PP. Trajectories of change in anxiety severity and impairment during and after treatment with evidence-based treatment for multiple anxiety disorders in primary care. Depress Anxiety. 2013 Nov;30(11):1099-106. doi: 10.1002/da.22149. Epub 2013 Jun 25. PMID 23801589
- [Result] Campbell-Sills L, Stein MB, Sherbourne CD, Craske MG, Sullivan G, Golinelli D, Lang AJ, Chavira DA, Bystritsky A, Rose RD, Welch SS, Kallenberg GA, Roy-Byrne P. Effects of medical comorbidity on anxiety treatment outcomes in primary care. Psychosom Med. 2013 Oct;75(8):713-20. doi: 10.1097/PSY.0b013e31829def54. Epub 2013 Jul 25. PMID 23886736
- [Result] Roy-Byrne P, Sullivan MD, Sherbourne CD, Golinelli D, Craske MG, Sullivan G, Stein MB. Effects of pain and prescription opioid use on outcomes in a collaborative care intervention for anxiety. Clin J Pain. 2013 Sep;29(9):800-6. doi: 10.1097/AJP.0b013e318278d475. PMID 23370069
- [Result] Bomyea J, Lang AJ, Craske MG, Chavira D, Sherbourne CD, Rose RD, Golinelli D, Campbell-Sills L, Welch SS, Sullivan G, Bystritsky A, Roy-Byrne P, Stein MB. Suicidal ideation and risk factors in primary care patients with anxiety disorders. Psychiatry Res. 2013 Aug 30;209(1):60-5. doi: 10.1016/j.psychres.2013.03.017. Epub 2013 Apr 19. PMID 23608160
- [Result] Glenn D, Golinelli D, Rose RD, Roy-Byrne P, Stein MB, Sullivan G, Bystritksy A, Sherbourne C, Craske MG. Who gets the most out of cognitive behavioral therapy for anxiety disorders? The role of treatment dose and patient engagement. J Consult Clin Psychol. 2013 Aug;81(4):639-649. doi: 10.1037/a0033403. Epub 2013 Jun 10. PMID 23750465
- [Result] Wetherell JL, Petkus AJ, Thorp SR, Stein MB, Chavira DA, Campbell-Sills L, Craske MG, Sherbourne C, Bystritsky A, Sullivan G, Roy-Byrne P. Age differences in treatment response to a collaborative care intervention for anxiety disorders. Br J Psychiatry. 2013 Jul;203(1):65-72. doi: 10.1192/bjp.bp.112.118547. Epub 2013 Apr 11. PMID 23580378
- [Result] Bomyea J, Lang AJ, Golinelli D, Craske MG, Chavira DA, Sherbourne CD, Rose RD, Campbell-Sills L, Welch SS, Sullivan G, Bystritsky A, Roy-Byrne P, Stein MB. Trauma Exposure in Anxious Primary Care Patients. J Psychopathol Behav Assess. 2013 Jun 1;35(2):254-263. doi: 10.1007/s10862-012-9327-0. PMID 23729989
- [Result] Niles AN, Sherbourne CD, Roy-Byrne PP, Stein MB, Sullivan G, Bystritsky A, Craske MG. Anxiety treatment improves physical functioning with oblique scoring of the SF-12 short form health survey. Gen Hosp Psychiatry. 2013 May-Jun;35(3):291-6. doi: 10.1016/j.genhosppsych.2012.12.004. Epub 2013 Jan 16. PMID 23332608
- [Result] Hunt J, Sullivan G, Chavira DA, Stein MB, Craske MG, Golinelli D, Roy-Byrne PP, Sherbourne CD. Race and beliefs about mental health treatment among anxious primary care patients. J Nerv Ment Dis. 2013 Mar;201(3):188-95. doi: 10.1097/NMD.0b013e3182845ad8. PMID 23407203
- [Result] Sullivan G, Sherbourne C, Chavira DA, Craske MG, Gollineli D, Han X, Rose RD, Bystritsky A, Stein MB, Roy-Byrne P. Does a quality improvement intervention for anxiety result in differential outcomes for lower-income patients? Am J Psychiatry. 2013 Feb;170(2):218-25. doi: 10.1176/appi.ajp.2012.12030375. PMID 23377641
- [Result] Brown LA, Craske MG, Glenn DE, Stein MB, Sullivan G, Sherbourne C, Bystritsky A, Welch SS, Campbell-Sills L, Lang A, Roy-Byrne P, Rose RD. CBT competence in novice therapists improves anxiety outcomes. Depress Anxiety. 2013 Feb;30(2):97-115. doi: 10.1002/da.22027. Epub 2012 Dec 5. PMID 23225338
- [Result] Zbozinek TD, Rose RD, Wolitzky-Taylor KB, Sherbourne C, Sullivan G, Stein MB, Roy-Byrne PP, Craske MG. Diagnostic overlap of generalized anxiety disorder and major depressive disorder in a primary care sample. Depress Anxiety. 2012 Dec;29(12):1065-71. doi: 10.1002/da.22026. Epub 2012 Nov 26. PMID 23184657
- [Result] Campbell-Sills L, Sherbourne CD, Roy-Byrne P, Craske MG, Sullivan G, Bystritsky A, Lang AJ, Chavira DA, Rose RD, Shaw Welch S, Stein MB. Effects of co-occurring depression on treatment for anxiety disorders: analysis of outcomes from a large primary care effectiveness trial. J Clin Psychiatry. 2012 Dec;73(12):1509-16. doi: 10.4088/JCP.12m07955. PMID 23290323
- [Result] Joesch JM, Sherbourne CD, Sullivan G, Stein MB, Craske MG, Roy-Byrne P. Incremental benefits and cost of coordinated anxiety learning and management for anxiety treatment in primary care. Psychol Med. 2012 Sep;42(9):1937-48. doi: 10.1017/S0033291711002893. Epub 2011 Dec 13. PMID 22152230
- [Result] Bystritsky A, Hovav S, Sherbourne C, Stein MB, Rose RD, Campbell-Sills L, Golinelli D, Sullivan G, Craske MG, Roy-Byrne PP. Use of complementary and alternative medicine in a large sample of anxiety patients. Psychosomatics. 2012 May-Jun;53(3):266-72. doi: 10.1016/j.psym.2011.11.009. Epub 2012 Feb 1. PMID 22304968
- [Result] Curran GM, Sullivan G, Mendel P, Craske MG, Sherbourne CD, Stein MB, McDaniel A, Roy-Byrne P. Implementation of the CALM intervention for anxiety disorders: a qualitative study. Implement Sci. 2012 Mar 9;7:1-11. doi: 10.1186/1748-5908-7-14. PMID 22404963
- [Result] Rose RD, Lang AJ, Welch SS, Campbell-Sills L, Chavira DA, Sullivan G, Sherbourne C, Bystritsky A, Stein MB, Roy-Byrne PP, Craske MG. Training primary care staff to deliver a computer-assisted cognitive-behavioral therapy program for anxiety disorders. Gen Hosp Psychiatry. 2011 Jul-Aug;33(4):336-42. doi: 10.1016/j.genhosppsych.2011.04.011. Epub 2011 Jun 8. PMID 21762829
- [Result] Stein MB, Roy-Byrne PP, Craske MG, Campbell-Sills L, Lang AJ, Golinelli D, Rose RD, Bystritsky A, Sullivan G, Sherbourne CD. Quality of and patient satisfaction with primary health care for anxiety disorders. J Clin Psychiatry. 2011 Jul;72(7):970-6. doi: 10.4088/JCP.09m05626blu. Epub 2011 Feb 22. PMID 21367351
- [Result] Craske MG, Stein MB, Sullivan G, Sherbourne C, Bystritsky A, Rose RD, Lang AJ, Welch S, Campbell-Sills L, Golinelli D, Roy-Byrne P. Disorder-specific impact of coordinated anxiety learning and management treatment for anxiety disorders in primary care. Arch Gen Psychiatry. 2011 Apr;68(4):378-88. doi: 10.1001/archgenpsychiatry.2011.25. PMID 21464362
- [Result] Sherbourne CD, Sullivan G, Craske MG, Roy-Byrne P, Golinelli D, Rose RD, Chavira DA, Bystritsky A, Stein MB. Functioning and disability levels in primary care out-patients with one or more anxiety disorders. Psychol Med. 2010 Dec;40(12):2059-68. doi: 10.1017/S0033291710000176. Epub 2010 Feb 11. PMID 20146834
- [Result] Roy-Byrne P, Craske MG, Sullivan G, Rose RD, Edlund MJ, Lang AJ, Bystritsky A, Welch SS, Chavira DA, Golinelli D, Campbell-Sills L, Sherbourne CD, Stein MB. Delivery of evidence-based treatment for multiple anxiety disorders in primary care: a randomized controlled trial. JAMA. 2010 May 19;303(19):1921-8. doi: 10.1001/jama.2010.608. PMID 20483968
- [Result] Chavira DA, Stein MB, Golinelli D, Sherbourne CD, Craske MG, Sullivan G, Bystritsky A, Roy-Byrne PP. Predictors of clinical improvement in a randomized effectiveness trial for primary care patients with panic disorder. J Nerv Ment Dis. 2009 Oct;197(10):715-21. doi: 10.1097/NMD.0b013e3181b97d4d. PMID 19829198
- [Result] Craske MG, Rose RD, Lang A, Welch SS, Campbell-Sills L, Sullivan G, Sherbourne C, Bystritsky A, Stein MB, Roy-Byrne PP. Computer-assisted delivery of cognitive behavioral therapy for anxiety disorders in primary-care settings. Depress Anxiety. 2009;26(3):235-42. doi: 10.1002/da.20542. PMID 19212970
- [Derived] Campbell-Sills L, Roy-Byrne PP, Craske MG, Bystritsky A, Sullivan G, Stein MB. Improving outcomes for patients with medication-resistant anxiety: effects of collaborative care with cognitive behavioral therapy. Depress Anxiety. 2016 Dec;33(12):1099-1106. doi: 10.1002/da.22574. Epub 2016 Oct 24. PMID 27775823
- [Derived] Jakubovski E, Bloch MH. Anxiety Disorder-Specific Predictors of Treatment Outcome in the Coordinated Anxiety Learning and Management (CALM) Trial. Psychiatr Q. 2016 Sep;87(3):445-64. doi: 10.1007/s11126-015-9399-6. PMID 26563229
- [Derived] Kelly JM, Jakubovski E, Bloch MH. Prognostic subgroups for remission and response in the Coordinated Anxiety Learning and Management (CALM) trial. J Clin Psychiatry. 2015 Mar;76(3):267-78. doi: 10.4088/JCP.13m08922. PMID 25562579

RESULTS

PARTICIPANT FLOW:
Groups:
- CALM Intervention: Participants assigned to coordinated anxiety learning and management (CALM)--
  CALM consists of: patient choice of Cognitive Behavioral Therapy (CBT), psychotropic (anti-anxiety) medication optimization or both.
  Optimization: 8 weeks of an evidence based anxiety medication at appropriate dose
  Cognitive-behavioral therapy: Participants in CALM will choose to receive CBT, medication, or both for the treatment of their anxiety. CBT includes computer-assisted CBT with an anxiety clinical specialist.
  Psychotropic medication optimization: For those participants in CALM who choose medication, the ACS will facilitate the delivery of, and adherence to, anti-anxiety medication which will be prescribed by the participants' PCP.
Period: Overall Study
Arm/Group | CALM Intervention | Treatment as Usual (TAU)
Started | 503 | 501
Completed | 409 | 395
Not Completed | 94 | 106
Not completed — Lost to Follow-up | 74 | 65
Not completed — Withdrawal by Subject | 18 | 38
Not completed — Death | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CALM Intervention | Treatment as Usual (TAU) | Total
Number analyzed (Participants) | 503 | 501 | 1004
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.3 (13.2) | 43.7 (13.7) | 43.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 359 | 355 | 714
  Male | 144 | 146 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 104 | 92 | 196
  Not Hispanic or Latino | 399 | 409 | 808
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 9
  Asian | 11 | 7 | 18
  Native Hawaiian or Other Pacific Islander | 2 | 2 | 4
  Black or African American | 40 | 57 | 97
  White | 333 | 331 | 664
  More than one race | 72 | 61 | 133
  Unknown or Not Reported | 40 | 39 | 79
Region of Enrollment [Number; unit: participants]
  United States | 503 | 501 | 1004

OUTCOME MEASURES:

1. Primary Outcome: BSI-12 (Anxiety and Somatization Subscales)
Description: 12 items from the Brief Symptom Inventory that measure anxiety and anxiety0related physical symptoms
Time Frame: Measured at Month 18
Measure: Number; unit: number of responders
Arm/Group | CALM Intervention | Treatment as Usual (TAU)
Number analyzed (Participants) | 503 | 501
number of responders | 325 | 258

2. Secondary Outcome: Functioning Outcomes as Measured by 3-item Sheehan Disability Scales and SF-12 and Disorder-specific Severity Scales as Measured by the ASI, PDSS-SR, GADS (Modified), SPIN, PCL-C, and the PHQ-9
Time Frame: Measured at Month 18
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 18 months
Description: As all treatments were part of standard care, both CBT and psychotropic medications routinely employed in clinical settings, no specific AE assessments were performed as would be done in clinical drug trials.
Arm/Group | CALM Intervention | Treatment as Usual (TAU)
All-Cause Mortality (participants affected / at risk) | 2/503 | 3/501
Serious Adverse Events (participants affected / at risk) | 0/503 | 0/501
Other Adverse Events (participants affected / at risk) | 0/503 | 0/501

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No